CLINICAL TRIAL: NCT00774280
Title: Randomized Comparison of Once-daily Intravenous Busulfan Plus Cyclophosphamide Versus Fludarabine as a Conditioning Regimen for Allogeneic Hematopoietic Cell Transplantation in Leukemia and Myelodysplastic Syndrome
Brief Title: Busulfan Plus Cyclophosphamide vs Fludarabine as a Conditioning Regimen
Acronym: BuCyvsBUFlu
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cooperative Study Group A for Hematology (Network)
Responsible Party: Je-Hwan Lee, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-005
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2011-02

CONDITIONS: Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ArmI(BuCy) (No Intervention): * Intravenous busulfan (Busulfex®; Orphan Medical, Minnetonka, MN) 3.2 ㎎/㎏ in normal saline 500 ㎖ i.v. over 3 hours on days -7 to -4
  * Cyclophosphamide 60 ㎎/㎏ in D5W 200 ㎖ i.v. over 1-2 hours on days -3 and -2
  Interventions: Drug: BuCy vs BuFlu
- Arm II (BuFlu) (No Intervention): * Intravenous busulfan 3.2 ㎎/㎏ in normal saline 500 ㎖ i.v. over 3 hours on days -7 to -4.
  * Fludarabine (Fludara®, Schering AG, Berlin, Germany) 30 ㎎/㎡ i.v. over 30 minutes in D5W 100 ㎖ on days -6 to -2
  Interventions: Drug: BuCy vs BuFlu

INTERVENTIONS:
Drug: BuCy vs BuFlu — Arm 1:BuCy Arm 2:BuFlu
  Other Names: busulfan plus cyclophosphamide versus fludarabine

SUMMARY:
1. At the same time of registration, patients will be randomized to one of the two conditioning therapy groups; Arm I (intravenous busulfan plus cyclophosphamide; BuCy) or Arm II (intravenous busulfan plus fludarabine; BuFlu).
2. Randomization will be a stratified permuted-block design. 2.1The patients will be stratified into standard risk vs. high risk group, and related vs. unrelated donor. Standard risk group will be defined as follows: patients with acute leukemia in first remission, CML in chronic phase, and MDS (RA or RARS categories). High risk group will be defined as follows: patients with acute leukemia in relapse or in second or subsequent remission, CML in accelerated or blastic phase, and MDS (CMMoL or RAEB categories).

2.2.Pre-assigned block size is 8.

DETAILED DESCRIPTION:
1. TREATMENT PLAN

   * The patients will be admitted to laminar air flow room.
   * The patients will have triple lumen Hickman central venous catheter (CVC) placed. Vancomycin 1 gm IV immediately prior to CVC placement and 1 gm q 12 hours for 3 doses. Chest X-ray should be taken after CVC placement to confirm the location of CVC and absence of pneumothorax.
   * Lumbar puncture will be done and intrathecal preservative free methotrexate 10 ㎎/㎡ (not to exceed 12 ㎎ total) will be given. Folinic acid 15 ㎎ will be given po or IV 24 hours after intrathecal methotrexate and q 6 hours for a total of 4 doses.
   * Menstruating women will be given norethindrone (Norlutate) 10 ㎎ po daily.
2. The preparatory regimen is as follows:

   * Conditioning therapy will start on day -7 in patients who are randomized to receive intravenous busulfan (Busulfex®; Orphan Medical, Minnetonka, MN) plus cyclophosphamide. Busulfex 3.2 ㎎/㎏ will be administered once daily for 4 days (days -7 to -4) followed by cyclophosphamide 60 ㎎/㎏ in D5W 200 ㎖ i.v. over 1-2 hours on days -3 and -2. Busulfex will be diluted in normal saline 500 ㎖ and infused over 3 hours by pump through a central venous catheter The doses of Busulfex and cyclophosphamide will be calculated using following guideline: 1) if actual body weight (ABW) of the patient is less or equal to ideal body weight (IBW), ABW will be used. 2) if ABW is greater than IBW but by less than 20%, then IBW will be used. 3) if ABW is greater than IBW by more or equal to 20 %, then the dose will be based on; IBW + 25 % (ABW-IBW). IBW is calculated as follows: 50 ㎏ + 2.3 ㎏ (Height in inch - 60) in male, and 45.5 ㎏ +2.3 ㎏ (Height in inch -60) (1 inch= 2.54 ㎝).
   * Conditioning therapy will start on day -7 in patients who are randomized to receive Busulfex plus fludarabine (Fludara®, Schering AG, Berlin, Germany). Busulfex 3.2 ㎎/㎏ will be administered once daily for 4 days (days -7 to -4) and fludarabine 30 ㎎/㎡ will be infused intravenously over 30 minutes in D5W 100 ㎖ for 5 consecutive days (days -6 to -2). The dose of Busulfex will be calculated using above-mentioned guideline (see 5.5.1). The dose of fludarabine will be calculated using ABW.
3. GVHD prophylaxis

   * All patients will receive cyclosporine 1.5 ㎎/㎏ in NS 100 ㎖ i.v. over 2-4 hours q 12 hrs (dose of cyclosporine rounded to nearest 5 ㎎) starting day -1 at 9 a.m. Cyclosporine dose will be adjusted to provide appropriate level and according to the change of renal function (see Appendix II).
   * When the patients can tolerate oral medications, cyclosporine can be given p.o. 3 ㎎/㎏ (or two times the i.v. dose) q 12 hrs.
   * Cyclosporine dose will be decreased by 10 % every month starting day 60 of BMT provided that there is no clinical evidence of GVHD.
   * In addition to cyclosporine, methotrexate 15 ㎎/㎡ will be given intravenously on day 1 and 10 ㎎/㎡ on days 3, 6, and 11. The dose of methotrexate will be decreased or omitted according to the guideline provided in Appendix III.
   * Methotrexate will not be given to patients with acute leukemia or MDS who will receive hematopoietic cell graft from an HLA-matched sibling donor
4. Bone marrow cell infusion

   * For ABO matched or minor mismatched transplantation, premedication with Avil 45.5mg I.v. push and tylenol 600 ㎎ p.o. will be given. Stem cell will be infused over 1-2 hrs.
   * For major ABO mismatched transplantation, premedication with Avil 45.5 ㎎ i.v. push, tylenol 600 ㎎ p.o., 10 % mannitol 100 g i.v. over 4 hrs will be started 30 min before stem cell infusion, and hydrocortisone 250 ㎎ i.v. will be given immediately before and 30 min of stem cell infusion.
5. Supportive cares.

   * Dilantin 15 ㎎/㎏ (ABW) in NS 200 ㎖ i.v. over 1 hour for loading on day -8, then 200 ㎎ p.o. bid through day -5. Dilantin dose should be adjusted to provide therapeutic level.
   * Allopurinol 300 ㎎/day p.o. qd day -8 to -2.
   * Nystatin powder to groin, axilla, and perianal area bid from day -8 until absolute neutrophil count (ANC) > 3,000/㎕.
   * Sodium bicarbonate/saline mouthwash qid until mucositis is resolved.
   * Fluconazole 100 ㎎/day p.o. qd until ANC > 3,000/㎕.
   * Ciprofloxacin 500 ㎎ p.o. bid (for selective bowel decontamination) until ANC > 3,000/㎕. With the first fever spike, ciprofloxacin will be discontinued and broad spectrum antibiotics will be begun.
   * Hydration will be done with 0.9 % NS at 100 ㎖/hour while the patients are receiving busulfan.
   * IV Immunoglobulin 500 ㎎/㎏ (ABW) i.v. over 6 hours every other week starting day -7 until day 120, then every month until day 180.
   * Prophylaxis against Herpes simplex virus will include acyclovir 250 ㎎/㎡ in D5W 100 ㎖ i.v. q 8 hours starting at day -7. When the patient can tolerate oral medication, acyclovir will be given 200 ㎎ p.o. tid until day 180.
   * Prophylaxis against Pneumocystis carinii will include Bactrim SS 2 tablets p.o. bid with folinic acid 7.5 ㎎ p.o. bid, 2 days weekly, starting after engraftment through day 360.
   * Amoxacillin 250 ㎎ p.o. bid starting at day 70 through day 360.
   * G-CSF administration.
   * Starting day 5, G-CSF 300 ㎍ in 100 ㎖ of D5W will be given i.v. over 3 hours daily until ANC > 3,000/㎕.
   * If ANC drops below 1,000/㎕, G-CSF administration will resume and continue until ANC > 3,000/㎕.
6. In patients with acute leukemia or CML in blastic crisis, intrathecal methotrexate administration will be resumed after the patient recovered platelet count to over 50,000/㎕. Methotrexate 10 ㎎/㎡ (not to exceed 12 ㎎ total) will be given intrathecally once every 2 weeks for three times (total four doses including one given before preparatory regimen). Folinic acid 15 ㎎ will be given p.o. or i.v. 24 hours after intrathecal methotrexate and q 6 hours for a total of 4 doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute leukemia, chronic myelogenous leukemia, myelodysplastic syndrome, and other hematologic malignancies.
* Patients should have an HLA-identical or one-locus mismatched sibling, family or unrelated donor.
* Patients should be 15 years of age or older, but younger than 70 years.

Exclusion Criteria:

* Patients have major illness or organ failure.
* Patients have a psychiatric disorder or mental deficiency severe as to make compliance with the treatment unlike, and making informed consent impossible.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2002-05; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
related toxicities of two different conditioning regimens, intravenous once-daily busulfan plus cyclophosphamide (BuCy) vs. fludarabine (BuFlu) for allogeneic hematopoietic cell transplantation (HCT) in leukemia and myelodysplastic syndrome | 8years

CONTACTS AND LOCATIONS:
Overall Officials: Je-Hwan Lee, Doctor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee JH, Joo YD, Kim H, Ryoo HM, Kim MK, Lee GW, Lee JH, Lee WS, Park JH, Bae SH, Hyun MS, Kim DY, Kim SD, Min YJ, Lee KH. Randomized trial of myeloablative conditioning regimens: busulfan plus cyclophosphamide versus busulfan plus fludarabine. J Clin Oncol. 2013 Feb 20;31(6):701-9. doi: 10.1200/JCO.2011.40.2362. Epub 2012 Nov 5. PMID 23129746
- See also: BuCy vs BuFlu — http://www.google.co.kr